CLINICAL TRIAL: NCT06358495
Title: Improving Sleep to Prevent Depression & Anxiety in Adolescents at High Risk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Hotchkiss Brain Institute, University of Calgary (Other)
Responsible Party: Principal Investigator, Daniel Kopala Sibley, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB24-0253
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Insomnia; Sleep Disturbance; Depressive Symptoms; Anxiety Symptoms
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Parasomnias; Depression; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either CBT for insomnia or TAU waitlist with a psychoeducational pamphlet about sleep hygiene.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be blinded to participants' assigned condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive-Behavioural Therapy Group (Experimental): Participants will receive a 6 week online Cognitive behavioural therapy for insomnia (CBT-I) evidence-based psychotherapeutic intervention that combines cognitive and behavioural principles. Their parents will also be invited to participant in 1 virtual psychoeducation session.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- Treatment as Usual waitlist with Psychoeducational Pamphlet (Active Comparator): Control group participants will receive a pamphlet providing information on sleep hygiene that matches the information in CBT-I arm (e.g., having a bedtime routine, maintaining a sleep schedule, avoiding exercise within several hours of bed, avoiding bright screens before bed). Otherwise, they will be encouraged to continue with treatment they are receiving, if any. After the 19 week follow-up assessment, participants have the option of receiving the digitized CBT-I intervention.
  Interventions: Other: Active Control

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — Digital CBT-I is an online, six-module, self-guided CBT-I intervention. It includes videos and read information on behavioral (e.g., stimulus control, relaxation) and cognitive (e.g., restructuring, reducing arousal, and problem-solving) techniques, as well as psychoeducation (e.g., sleep hygiene). Participants complete homework following each session and track their sleep using an online diary. Young people could choose to involve their parents, for example, through completing sessions together. However, we will add a virtual session for parents as their involvement may improve adolescent engagement with the intervention as well as outcomes for adolescent sleep problems (Gradisar et al., 2011). This module will include an overview of the program components (behavioural, cognitive, and educational), goals and homework, and addresses parents' beliefs about sleep.
  Arms: Cognitive-Behavioural Therapy Group
Other: Active Control — Participants are encouraged to continue any care they are already receiving and will be placed on a wait-list for digital CBT-I after their final assessment. All activities participants try for improving their own sleep problems between assessments will be recorded and coded for.
  Arms: Treatment as Usual waitlist with Psychoeducational Pamphlet

SUMMARY:
Emerging evidence has shown that sleep interventions such as Cognitive Behavioral Therapy for Insomnia (CBT-I) improve depressive and anxiety symptoms in adults, even when the intervention is brief, such as four to six sessions. The overarching aim of the proposed research is to conduct a pilot trial to evaluate whether a brief intervention for insomnia adapted for improves sleep and subthreshold depressive and anxiety symptoms in adolescents at risk (i.e., with a parental history of depressive or anxiety disorders).

DETAILED DESCRIPTION:
A substantial body of literature has linked poor sleep or insomnia to the development of internalizing (i.e., depression and anxiety) disorders in adolescents. Emerging evidence has also shown that sleep interventions such as Cognitive Behavioral Therapy for Insomnia (CBT-I) substantially improve depressive and anxiety symptoms in adults, even when the intervention is brief, such as four to six sessions. However, no research has examined whether sleep interventions may be effective in preventing first lifetime onsets of internalizing disorders in adolescents at high risk of internalizing disorders, but who have yet to develop them. The overarching aim of the proposed research is to conduct a pilot trial to evaluate whether a brief intervention for insomnia adapted for adolescents improves sleep and subthreshold internalizing symptoms in high-risk adolescents. Results of this project would provide crucial preliminary evidence that a non-invasive, economical, and easily administered sleep-based intervention may prevent first onsets of the most common and debilitating illnesses in teens.

Among adolescents, internalizing disorders are a leading cause of global burden of disability, and unfortunately one of the leading causes of death due to suicide. Children with a parental history of internalizing disorders are 3-7 times more likely to develop internalizing disorders relative to children with no such family history. Approximately 75% of internalizing disorder onsets occur in adolescence. Affected youth are at risk for several sequelae including substance dependence, educational underachievement, and unemployment. For the majority of those who have had one episode, the disorder will become chronic. With each recurrence, treatment prognosis worsens. There is thus a critical need to prevent first lifetime onsets of internalizing disorders, among high-risk adolescents in particular, through interventions targeting modifiable risk factors. Improving sleep may be a feasible, economic, and effective method for prevention of internalizing disorders in high-risk teens.

Research Aims:

1. To examine if brief web-based CBT-I reduces insomnia symptoms and improves sleep quality in teens at risk for internalizing disorders, compared to a treatment as usual (TAU) waitlist group who receive a psychoeducational pamphlet about sleep hygiene.
2. To examine if CBT-I improves subthreshold internalizing symptoms in teens who have a family history of depressive or anxiety disorders but no clinically significant history themselves.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 12 and 18.
* Having at least one parent with a history of depressive or anxiety disorders but having no clinically significant history (per the Diagnostic and Statistical Manual of Mental Disorders 5) of internalizing disorders themselves.
* Adolescents who score 10/25 or greater on the Insomnia Severity Index, indicating subthreshold insomnia or greater.

Exclusion Criteria:

* Experiencing symptoms of sleep disorders other than insomnia (i.e. restless legs syndrome [RLS], sleep-disordered breathing [SDB].
* Having a history of untreated, serious psychiatric illness (i.e., bipolar disorder, schizophrenia).
* Active suicidal ideation.
* Currently taking prescribed medications for sleep problems.
* Moderate to severe head injury.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index | Change between 3 time-points: baseline, 7-week follow-up, 19-week follow-up.
  The ISI is a 7-item questionnaire designed to identify cases of insomnia and evaluate treatment outcomes. The ISI assesses severity of sleep onset, sleep maintenance and early wakening problems, sleep dissatisfaction, and perceived distress caused by sleep problems. It was found to be a clinically useful tool in assessing changes in insomnia symptoms and had been reliably used in treatment research with adolescents. Scores on the ISI range from 0-28 with higher scores indicating greater insomnia severity.
Pittsburgh Sleep Quality Index | Change between 3 time-points: baseline, 7-week follow-up, 19-week follow-up.
  The PSQI instrument is used in assessing one's sleep quality during the previous month. It consists of 19 self-rated items. It has been reliably used in treatment research with adolescents. Scores range from 0 to 19, with higher scores indicating worse sleep quality.
Internalizing Symptoms Subscale of the Youth Self-Report | Change between 3 time-points: baseline, 7-week follow-up, 19-week follow-up.
  The internalizing symptoms subscale of the Youth Self Report (YSR) questionnaire is a widely used measure of global internalizing (depression, anxiety, and somatic) symptoms. T-scores which range from 26 to 100 are generated, with higher scores indicating greater symptom severity.

SECONDARY OUTCOMES:
Sleep Logs - Total sleep time | Change between 3 time-points: baseline, 7-week follow-up, 19-week follow-up.
  Sleep logs provide self-reported subjective sleep. Participants will be asked to report on their estimated total sleep time.
Sleep Logs - Onset latency | Change between 3 time-points: baseline, 7-week follow-up, 19-week follow-up.
  Sleep logs provide self-reported subjective sleep. One of the variables participants will report is the amount of time they think it takes them to fall asleep.
Sleep Logs - Wake after sleep onset | Change between 3 time-points: baseline, 7-week follow-up, 19-week follow-up.
  Sleep logs provide self-reported subjective sleep. One of the variables participants will report is the amount of time they think they spent awake at night after initially falling asleep.
Sleep Logs - Sleep efficiency | Change between 3 time-points: baseline, 7-week follow-up, 19-week follow-up.
  Sleep logs provide self-reported subjective sleep. Sleep efficiency (percent of time spent asleep while in bed) will be calculated based on participants reports of total sleep time divided by time spent in bed.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Kopala-Sibley, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Recognizing the importance of sharing results, data will be shared in accordance with the International Committee of Medical Journal Editors' guidelines, which state that authors can share with others the deidentified individual participant data underlying results presented in the trial reports (including tables, figures, and appendices or supplementary material) no later than 6 months after publication. Data will be made available upon request to the primary investigator.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data can be shared no later than 6 months after publication, and will be available until study records are destroyed in accordance with research ethics board requirements (min 10 years post collection).